CLINICAL TRIAL: NCT04285957
Title: Italian Translation and Transcultural Validation of Two Assessment Tools for Participation in Stroke Survivors: the Frenchay Activity Index and the Walking Handicap Classification (FAIWHC)
Brief Title: Italian Translation and Transcultural Validation of Frenchay Activity Index and Walking Handicap Classification in Stroke
Acronym: FAIWHC
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: FAIWHC
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Stroke Sequelae
Keywords: participation; Frenchay Activity Index; Walking Handicap Classification; Stroke Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-test Group: Consecutive recruitment of 10 post-stroke patients undergoing intensive rehabilitation treatment at the Neurological Rehabilitation Unit, Foundation don Gnocchi Scientific Institute.
  Inclusion criteria: age 18-90, stroke occurred within 3 months from enrollment; clinical stability (SIC = 0). The exclusion criteria are: stroke recurrence; visual and / or hearing disorders; cognitive decline (MMSE <21) and/or severe aphasia, which would limit the the patients' understanding of and the reliable answering to the two assessment tools
  Interventions: Other: Questionnaire administration pre test
- Validation Group: Recruitment of 60 post-stroke patients undergoing intensive rehabilitation treatment at the Neurological Rehabilitation Unit, Foundation don Gnocchi Scientific Institute.Inclusion criteria: age 18-90, stroke occurred within 8 months from enrollment; clinical stability (SIC = 0). If the following criteria are present: visual and / or hearing disorders; cognitive decline (MMSE <21) and/or severe aphasia, which would limit the patients' understanding of and the reliable answering to the two assessment tools, the interview shall be carried out with a proxy
  Interventions: Other: Questionnaire administration - validation

INTERVENTIONS:
Other: Questionnaire administration pre test — Pre-test:
  Two expert physicians/physical therapist shall be involved in the questionnaire administration (A/B). The questionnaires shall be randomly administered to the patients by one operator at T0 the same test shall be readministered after 1-2 weeks by another operator (T1), blind to the first assessment; the second operator shall also administer the additional measures (SIP and RMI);
  Other Names: Questionnaire administration - validation
  Groups: pre-test Group
Other: Questionnaire administration - validation — Validation Two expert physicians shall be involved in the questionnaire administration (A/B). The questionnaires shall be randomly administered to the patients by one operator at T0 the same test shall be readministered after 1-2 weeks by another operator (T1), blind to the first assessment; the second operator shall also administer the additional measures (SIP and RMI); In case the patient is unable to be interviewed due to aphasia cognitive or sensorial problems, a proxy would be interviewed both at T0 and at T1 (the same proxy would be interviewed both times)
  Groups: Validation Group

SUMMARY:
This study is aimed at providing an Italian version of two assessment tools for participation in stroke patients, the Frenchay Activity Index (FAI) and the Walking Handicap Classification (WHC) by a standardized translation and transcultural validation protocol. The protocol includes a pre-test of the Italian version on ten patients, a final revision, and a validation on a sample of 60 stroke patients.

DETAILED DESCRIPTION:
This study is aimed at providing an Italian version of two tools to assess participation in stroke patients, the Frenchay Activity Index (FAI) and the Walking Handicap Classification (WHC). These tools have been recently indicated for the assessment of participation in Stroke patients by the Italian Association of Physical and Rehabilitation Medicine (Minimal Stroke Assessment Protocol - PMIC2); they are currently used in Italian research and clinical settings, but no official translation exists. The process requires a standardized translation protocol, including forward and backward translation, using a multistep revision structure, to ensure conceptual and semantic equivalence. The validation process includes a pilot evaluation of on 10 individuals post-stroke admitted to the Neurological Rehabilitation Unit, Foundation Don Gnocchi Scientific Institute, and a validation on a sample of 60 stroke patients including reliability, internal consistency and concurrent validity assessment of the translated version against the Sickness Impact Profile (SIP) - Italian version and the Rivermead Mobility Index (RMI) - Italian version, respectively

ELIGIBILITY:
Pre-test: consecutive recruitment of 10 post-stroke patients undergoing intensive rehabilitation treatment at the Neurological Rehabilitation Unit, Foundation don Gnocchi Scientific Institute.

Inclusion criteria:

* age 18-90;
* stroke occurred within 3 months from enrollment;
* clinical stability (SIC = 0).

Exclusion criteria:

* stroke recurrence;
* visual and / or hearing disorders;
* cognitive decline (MMSE <21) and/or severe aphasia, which would limit the the patients' understanding of and the reliable answering to the two assessment tools

Validation: recruitment of 60 post-stroke patients undergoing intensive rehabilitation treatment at the Neurological Rehabilitation Unit, Foundation don Gnocchi Scientific Institute-

Inclusion criteria:

* age 18-90,
* stroke occurred within 8 months from enrollment;
* clinical stability (SIC = 0).

Criteria for carrying out the interview with a proxy. If a proxy is not available, the patient is excluded:

* visual and / or hearing disorders;
* cognitive decline (MMSE <21) and/or severe aphasia, which would limit the patients' understanding of and the reliable answering to the two assessment tools.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-test: 10 consecutively recruited post-stroke patients undergoing intensive rehabilitation treatment at the Neurological Rehabilitation Unit, Foundation don Gnocchi Scientific Institute.Inclusion and exclusion criteria listed in the dedicated section.
  Validation: 60 post-stroke patients undergoing intensive rehabilitation treatment at the Neurological Rehabilitation Unit, Foundation don Gnocchi Scientific Institue.Inclusion and exclusion criteria listed in the dedicated section. If the following are present: visual and / or hearing disorders; cognitive decline (MMSE <21) and/or severe aphasia, which would limit the patients' understanding of and the reliable answering to the two assessment tools, the interview shall be carried out with a proxy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Interrater reliability | 1 year
  Intraclass Correlation Coefficient >=0,70
Internal consistency (FAI) | 1 year
  Cronbach's alpha>=0,70
concurrent validity of FAI against SIP | 1 year
  Spearman's coefficient >=0.25-0.50
concurrent validity of WHC against RMI | 1 year
  Spearman's coefficient >=0.25-0.50

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Cecchi, Md, Principal Investigator — Fondazione don Carlo Gnocchi IRCCS
Locations (1):
- Fondazione don Gnocchi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided